CLINICAL TRIAL: NCT00790491
Title: Automated Guidance Tool for Medical Encounters Addressing Therapeutic Lifestyle Changes (AuGMEnT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: Viocare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007-11
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Heart Disease; Diabetes
Keywords: reduction in risk of heart disease and diabetes
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: guidance tool for providers for lifestyle changes

INTERVENTIONS:
Behavioral: guidance tool for providers for lifestyle changes — automated guidance tool for medical providers involved in patient encounters addressing lifestyle changes. Addresses dietary and physical activity. Seeks to reduce cardiac disease risk.

SUMMARY:
ABSTRACT Although most primary healthcare practitioners recognize the important relationship among nutrition, physical activity and health, few incorporate either dietary or physical activity counseling into routine practice. AUGMENT will employ interactive technology to support effective patient life-style counseling during routine office visits. AUGMENT technology will automate the administration, collection, and analysis of dietary and physical activity questionnaires, and it will guide counseling and present intervention resources and strategies tailored to the patient's unique needs. Using tablet computers, wireless LANs, and inexpensive Internet communications, AUGMENT will have advantages over existing tools: 1.) Lower usage costs (minimal office personal required), 2.) Ability to customize the system, and 3.) Real-time, comprehensive assessment.

The AUGMENT system efficiently and relentlessly gathers important healthcare information (such as total fat, type of fat consumption; fruit and vegetable consumption; fiber and micronutrient intake; and energy output). This means patients are less likely to have their preventive needs overlooked by a busy practitioner. The assessment includes questions to determine the amount of effort the patient will commit to improved health. This will enable the physician to effectively guide the patient via targeted recommendations, obtainable goals, and a course of action that is both preventive and prescriptive; and to monitor progress. Patients who receive objective assessments of their healthcare practices and recommendations based on their own unique health history will be more likely to accept and act on the recommendations.

The specific aims of the study are to: 1) Incorporate key elements of a previously developed prototype tool into a dietary and physical activity risk assessment system, 2) Create a provider training tool to build proficiency in using AUGMENT for counseling to reduce disease risk.

3) Validate the AUGMENT dietary and physical activity assessments using dietary recalls and accelerometer data, 4) Complete a process evaluation of the AUGMENT program by using it in interventions managed by six physicians with at least 240 patients, and 5) Survey participating providers and patients to assess acceptability of AUGMENT within a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* adult patients at Staywell Community Health Center, Waterbury CT

Exclusion Criteria:

* terminally ill
* pregnant women
* children
* decisionally impaired / dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Validate the AUGMENT dietary and physical activity assessments using dietary recalls and accelerometer data, | 2 years

SECONDARY OUTCOMES:
Survey participating providers and patients to assess acceptability of AUGMENT within a clinical setting. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Waterbury Management Resources and Family Care, Waterbury, Connecticut, United States